CLINICAL TRIAL: NCT03013855
Title: Efficacy of Fecal Immunochemical Test Using Digital Rectal Exam
Acronym: FIT-DRE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-34258
Record Dates: First submitted 2016-08-17; First posted 2017-01-09 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Fecal Immunochemical Test
Keywords: Digital rectal exam; Colon cancer screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- FIT-SOC (Active Comparator): Fecal immunochemical test performed on spontaneously passed stool as noted in the standard instructions.
  Interventions: Device: FIT-SOC
- FIT-DRE (Experimental): Fecal immunochemical test completed with stool collected during digital rectal exam.
  Interventions: Device: FIT-DRE

INTERVENTIONS:
Device: FIT-SOC — Study subjects will be given a standard kit for fecal immunochemical test by their primary healthcare provider. As per standard practice, the patient will take the kit home and use the included FIT applicator to collect a stool sample from spontaneously passed stool during a regular bowel movement. The patient will then mail the stool sample to the lab in a pre-paid envelope, which is provided in the kit.
  Arms: FIT-SOC
Device: FIT-DRE — Study subjects will have a digital rectal exam completed by their primary care providers during the physical exam portion of a routine clinic visit. The stool collected on the examiner's finger will be applied to the FIT applicator in the standard kit, which will then be sent to the lab for processing.
  Arms: FIT-DRE

SUMMARY:
This study will investigate the use of digital rectal exam (DRE) to obtain stool samples for the fecal immunochemical test (FIT) in patients due for screening colonoscopy and in pre-operative patients with known colorectal cancer. FIT is currently FDA-approved for spontaneous stool and DRE, however, samples are not commonly obtained by DRE. In addition, some clinicians remain skeptical about the accuracy of FIT using stool obtained from DRE. This study aims to assess the correlation between FIT using the stool sample from DRE (FIT-DRE) and standard of care FIT (FIT-SOC). If good correlation is shown, the investigators may be able to demonstrate efficacy of FIT using a DRE in the clinic setting. This may help avoid logistical barriers, as well as improve compliance and adherence to colon cancer screening in the outpatient setting, eventually leading to improved quality of care.

DETAILED DESCRIPTION:
Fecal immunochemical testing (FIT) is an FDA-approved stool-based screening test for colorectal cancer. It offers a less invasive colorectal cancer screening option for patients who are not agreeable to colonoscopy and measures the level of Ab-globin complexes in the stool without direct interference with diet or medications. FIT has been shown to be selective for colorectal bleeding, as globin from the upper GI tract is digested by proteolytic enzymes. A meta-analysis of studies analyzing FIT showed a pooled sensitivity of 0.79 (95% CI 0.69-0.86) and specificity was 0.94 (CI 0.92-0.95). In a large study comparing FIT with another stool-based screening test, gFOBT, sensitivity of FIT was found to be 0.53-0.73 for CRC and 0.20-0.25 for advanced neoplasia compared to gFOBT, which showed 33.3% for CRC and 8.6% for advanced neoplasia. In addition, FIT requires fewer stool samples and the lack of dietary or medication modifications. As a result, compliance is likely to be higher, which is crucial for cancer detection.

A challenge inherent to stool-based screening tests is compliance with sample submission by the patients. FIT is meant to improve logistical barriers to screening because only one sample is needed, however, compliance rates with standard of care FIT (FIT-SOC) is approximately 50%. FIT using stool from a digital rectal exam (DRE) performed during a clinic visit may be an effective screening tool for patients preferring stool-based screening. FIT has been FDA-approved for the testing of spontaneously passed stool, as well as stool collected by DRE. Manufacturers of FIT have claimed that DRE provides a sufficient amount of stool for sampling, however, there are no validated studies to our knowledge which demonstrate adequate efficacy. As a result, FIT using DRE is not commonly done in clinical practice. This study aims to assess the correlation of FIT using DRE (FIT-DRE) with standard of care FIT (FIT-SOC) as a method of obtaining stool samples.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 50-75 who are due for colon cancer screening and scheduled for colonoscopy
* Preoperative patients with established diagnosis of colon cancer

Exclusion Criteria:

* Patients with a diagnosis of Inflammatory Bowel Disease (IBD).
* Patients who are pregnant.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Concordance between standard FIT results and DRE FIT results. | 1 year
  For example, the percentage of positive standard FIT results that also have positive DRE FIT results, and the percentage of negative standard FIT results that also have negative DRE FIT results.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jacobson, MD, Study Director — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee JK, Liles EG, Bent S, Levin TR, Corley DA. Accuracy of fecal immunochemical tests for colorectal cancer: systematic review and meta-analysis. Ann Intern Med. 2014 Feb 4;160(3):171. doi: 10.7326/M13-1484. PMID 24658694
- [Background] Brenner H, Tao S. Superior diagnostic performance of faecal immunochemical tests for haemoglobin in a head-to-head comparison with guaiac based faecal occult blood test among 2235 participants of screening colonoscopy. Eur J Cancer. 2013 Sep;49(14):3049-54. doi: 10.1016/j.ejca.2013.04.023. Epub 2013 May 22. PMID 23706981